CLINICAL TRIAL: NCT06639477
Title: Multi-site Randomized Controlled Trial Comparing the Efficacy of Behavioral Approaches to Improve Mood and Sleep in Adults
Brief Title: Assessing Improvements in Mood and Sleep Trial
Acronym: AIMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Emory University (Other); University of California, Berkeley (Other); University of California, Los Angeles (Other); Augusta University (Other); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen Smagula, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY24030049; R01MH137185 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Depression; Suicidality; Sleep
Keywords: Older Adults; Depression
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concealed Control Intervention (Active Comparator): Participants receive eight ~40 minute sessions (one per week) with a therapist/health coach. Specific information regarding the nature of the interventions is withheld to protect the scientific integrity of the study design.
  Interventions: Other: Treatment As Usual; Behavioral: Active Comparator
- Active Condition (Experimental): Participants receive eight ~40 minute sessions (one per week) with a therapist/health coach. Specific information regarding the nature of the interventions is withheld to protect the scientific integrity of the study design.
  Interventions: Other: Treatment As Usual; Behavioral: Active Condition

INTERVENTIONS:
Other: Treatment As Usual — In this trial, all participants will have depression symptoms and will be receiving TAU from their own doctors.
Behavioral: Active Condition — Participants receive eight ~40 minute sessions (one per week) with a therapist/health coach. Specific information regarding the nature of the interventions is withheld to protect the scientific integrity of the study design.
  Arms: Active Condition
Behavioral: Active Comparator — Participants receive eight ~40 minute sessions (one per week) with a therapist/health coach. Specific information regarding the nature of the interventions is withheld to protect the scientific integrity of the study design.
  Arms: Concealed Control Intervention

SUMMARY:
This is a multi-site randomized control trial involving people age 55+ years who have current depression symptoms plus another suicide risk indicator (either current suicidal ideation or a past history of attempt). Our goal is evaluate which of two different approaches works best to improve things like trouble sleeping, bad moods, and any suicidality.

Participants will complete diagnostic interviews, self-report scales, and wear an actigraphy device for the 8 weeks starting at the baseline visit.

DETAILED DESCRIPTION:
The main purpose of the study is to compare the effects of two approaches on sleep and mood including any symptoms of depression and suicidality. There will be 420 people invited to participate across three sites in the United States (University of Pittsburgh, UCLA, Augusta).

Participants will be randomized to receive one of two evidence-based programs that are designed to help improve outcomes. Each group will contain 210 participants. Researchers will enroll a total of 140 participants (70 in each group) at the University of Pittsburgh. Both groups will meet with a study therapist once a week to complete the assigned 8-week program. To determine which (if any) program has beneficial effect over time, researchers will ask participants to complete assessments of their sleep, mood, and health before and after the therapy. Certain information regarding the nature of the interventions is withheld to protect the scientific integrity of the study design.

There are three main study visits where participants will complete assessments about their sleep, mood, cognition and health. These would be:

* Before the therapy program begins
* Right after it ends
* Six months later

Around the time of each visit, researchers will ask participants to wear an actigraphy watch on their wrist 24/7 for a week while completing a sleep diary. The actigraphy watch is a wrist-watch like device that measures movement so that researchers can estimate the participant's activity and sleep levels.

After the first main visit is complete, participants will be randomly assigned to one of two programs that include meeting with a study clinician for 30-50 minutes each week for 8 weeks (8 sessions total). Both groups will receive educational information and, depending on the group the participants are assigned to, may include guided discussions, activities, and/or support addressing any stressors participants face, sleep problems, and/or depression.

During the therapy period, researchers would ask participants to continue wearing the actigraphy watch. Researchers would also ask participants to answer questions on the phone with study staff weekly (that would take about 30-40 minutes a week).

After the participant's last therapy session, researchers would repeat the phone assessments once a month until the last main visit occurs (six-months after therapy ends).

ELIGIBILITY:
Inclusion Criteria:

* Age 55 Years and older
* Patient Health Questionnaire -9 score of 10 or higher
* Past month Scale for Suicide Ideation score of 3 or higher OR any history of suicide attempt
* PROMIS Sleep Disturbance or impairment scale t-scores of 55 or higher
* Pharmacotherapy for depression meeting minimum adequate dose level as defined by FDA approval documents for at least 4 weeks.

Exclusion Criteria:

* Active suicide planning with intent or clinical judgement that suicide risk is too high for outpatient treatment OR being currently treated at an inpatient unit.
* Bipolar disorder
* Psychotic disorder
* Borderline personality disorder.
* Active Cognitive/Behavioral Therapy (e.g., CBT-I), current or upcoming esketamine (ketamine) treatment, or active phase of ECT/TMS treatment course.
* Illness with life expectancy of less than 1 year or plans to leave the study area
* Incapacity to consent/dementia diagnosis
* Active substance use disorder of at least moderate severity
* Active night-shift work

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Depression Symptom Response | six months post-treatment
  The outcome is the rate of clinically significant depression symptom responses six-months post treatment, defined as having ≥50% reduction in pre-treatment depression severity six-months posttreatment. Depression severity will be assessed as total scores from the 14 non-sleep items of the clinician rated GRID Hamilton Depression Rating Scale. Lower scores on the GRID Hamilton would indicate a reduction in depression symptoms.

SECONDARY OUTCOMES:
Change in Suicide Ideation Severity | from Enrollment to the end of treatment at 6-months post-intervention
  Measuring rates of clinically significant past-month active SI at the six-month follow-up defined as Columbia Suicide Severity Rating Scale (CSSR) ideation dimension scores ≥ 3. This level on the CSSR, equivalent to having at least SI with a method, was identified as an optimal cut-off for predicting future suicide death. Lower scores on the Columbia Suicide Severity Rating Scale would indicate lower levels of suicide ideation.
Suicide Behavior Outcomes | from Enrollment to the end of treatment at 6-months post-intervention
  Any suicidal behaviors over the six-month follow-up defined as escalating planning, suicide attempt, or suicide-related hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F Smagula, Ph.D, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - The Regents of the University of California, Los Angeles, Los Angeles, California
  - Augusta University, Augusta, Georgia
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the main measures of this study as reported in publications after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 5 years after article publication
Access Criteria: Researchers who provide methodologically sound proposal